CLINICAL TRIAL: NCT06058169
Title: Pilot Investigation on the Effects of Sub Acute (12 Week) Home Base Whole-body Vibration Training in Osteoarthritis.
Brief Title: Effects of Home Base Whole-body Vibration in Osteoarthritis. (VIBE-Rx2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2054289
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Whole Body Vibration; Osteo Arthritis Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Body Training (12 week) (Experimental)
  Interventions: Device: Sub Acute Whole Body Vibration Training

INTERVENTIONS:
Device: Sub Acute Whole Body Vibration Training — Participants will be given a personal vibration plate (equipped with stabilizing bars) to take home for training which will last for up 12 weeks. For this test the participant will be asked to stand on a vibration plate for up to 20 minutes. Participants will be instructed to remove any footwear and stand mid-center on the platform in a standing position with feet shoulder width apart. The participant will be asked to step on and off of the vibration plate. During the first four weeks, participants will be asked to complete 5-10 minutes of WBV per day, at least 4-5 days per week. At least 24 hours will be recommended in between sessions during weeks 1-4. Beginning at week 5, participants will be asked to increase WBV time to up to 15 minutes and/or reduce the duration of rest. Beginning at week 9, based on how the participant feels, the study team may adjust the WBV time/duration up to 20 minutes per session, 4-5 days per week.

SUMMARY:
The purpose of this proposal is to understand how the Vibrant Health Ultimate whole-body vibration (WBV) machine affects pain and inflammation in older adults. The investigators' hypothesize that sub-acute (12 weeks) WBV will lead to improvement in the level of knee pain and improve vascular function via a decrease in systemic inflammation.

DETAILED DESCRIPTION:
Knee osteoarthritis (KO) is a leading cause of disability and medical cost. Whole body vibration (WBV) has emerged as an exercise alternative that may be more tolerable than traditional forms of exercise, such as treadmill walking/running or cycling. Similar to traditional exercise, research supports that WBV can be very beneficial for your health. In fact, a single bout of WBV increases circulating concentrations of inflammatory markers. WBV is safe and effective, WBV training has been conducted in obesity, elderly, patients with diabetes, patients with lung disease, as well as patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Osteoarthritic knee pain for at least 6 months.
* Mean and women
* Ages 40-75 years old

Exclusion Criteria:

* <40 years old or >75 years old
* History of balance issues
* History of falls
* Epilepsy
* Pregnancy
* The use of whole-body vibration in the past 6 months
* Previous knee surgery within last 3 years
* Unable to stand for at least 20 minutes (for whole body vibration training)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Pressure Threshold assessed using the Jtech Medical Echo Algometer | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  change from baseline pain pressure threshold at 12 weeks. Pain Pressure Threshold (PPT) will be assessed using the Jtech Medical Echo Algometer. PPT is used to measure deep muscular tissue sensitivity. The test determines the amount of pressure over a given area in which a steadily increasing non-painful pressure stimulus turns into an uncomfortable or painful pressure sensation. The subject will lie supine. An investigator will assess PPT at the following sites: a) 2 cm below the medial edge of the patella and b) 2 cm below the lateral edge of the patella. Using the 1 cm2 probe, the investigator will place it perpendicular to each site and apply pressure at a rate of 0.5 kg/cm2/s. Each trial will stop when the subject reports pain. The investigator will take 3 trials at each site; the average of the 3 trials, recorded in kg/cm2, will be used for statistical analysis.

SECONDARY OUTCOMES:
Change in Pulse Wave Velocity (PWV) | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  Change from baseline PWV at 12 weeks. Measured by Shygmocor Xcel in m/s.
Change in IL-6 | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  change from baseline concentrations of Interleukin 6 (IL-6) obtained via blood draw at 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University/Georgia Prevention Institute/ Laboratory of Integrative and Exercise Physiology, Augusta, Georgia, United States